CLINICAL TRIAL: NCT01278771
Title: Coronary Anomalies in Congenital Heart Disease
Acronym: CHD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Avraham Lorber MD, Rambam Medical Center, Meyer Children's Hospital
Other Study IDs: 0496CTIL
Record Dates: First submitted 2011-01-16; First posted 2011-01-19 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2010-10

CONDITIONS: Congenital Heart Disease
Keywords: CHD
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective study. The investigators shall review the angiography data of 1200 consecutive cardiac catheterizations of children and babies with CHD (Congenital Heart Disease) since 1998 till now.

Coronary artery origin and course will be evaluated in relation to the morphologic cardiac anomalies.

Coronary artery anomalies will be described and statistical analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* cradiac catheterization with angiography with congenital heart disease.

Exclusion Criteria:

* no congenital heart disease.

Max Age: 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1200 patients with Congenital Heart Disease who underwent Cardiac catheterization with angiography.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2011-03

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Lorber, Prof, Principal Investigator — Rambam Medical Health Care Campus